CLINICAL TRIAL: NCT04372095
Title: Androcur® (Cyproterone Acetate) and Meningioma Development: a Genotype-environment Association Study
Acronym: ANDROMEDE-F
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200222; 2020-A00045-34 (Registry Identifier: IDRCB)
Record Dates: First submitted 2020-04-30; First posted 2020-05-01 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Meningioma
Keywords: meningioma; predisposition; genetic
MeSH Terms: conditions — Meningioma; Disease Susceptibility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Oral smears: the sampling of oral smears will be collected by subjects themselves at home and sent to the Biological Research Center (CRB) of Neuro-Oncothèque of La Pitie Salpêtrière hospital. Each sampling will be accompanied by an inform consent signed by the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- group 1: Exposed to CPA + Meningioma: Meningioma diagnosed in women by medical imaging examination and confirmed histologically if surgery is performed.
  Cyproterone acetate taken for at least 6 months.
  Interventions: Procedure: oral smears
- group 2: Exposed to CPA without Meningioma: Women exposed to Cyproterone acetate without developing any meningioma Absence of meningioma assessed by a normal cerebral MRI . Cyproterone acetate taken for at least 5 years.
  Interventions: Procedure: oral smears
- group 3: Not exposed to CPA, Meningioma diagnosed: Meningioma in women not exposed to cyproterone acetate. Meningioma diagnosed by medical imaging examination and confirmed histologically if surgery was necessary.
  Never exposed to cyproterone acetate.
- group 4: General population: Subjects (women) never diagnosed with meningioma and not exposed to cyproterone acetate.

INTERVENTIONS:
Procedure: oral smears — oral smears
  Groups: group 1: Exposed to CPA + Meningioma; group 2: Exposed to CPA without Meningioma

SUMMARY:
The primary objective of the study is to create a biobank of oral smears permitting to identify the genetic locus/loci associated with an increased risk to develop meningiomas after cyproterone acetate (CPA) (Androcur®) treatment, using a GWAS approach.

As the secondary objectives, the study aims:

* to evaluate the importance of the genetic susceptibility.
* to record the frequence of homonodependant cancers occuring in female patients with Androcur® associated meningioma and in their first-degree relatives.
* to describe clinical, radiological, histological characteristics of the patients who have developed meningioma after cyproterone acetate exposure.

DETAILED DESCRIPTION:
The increased risk to develop a meningioma has recently been established for patients received the cyproterone acetate.

The investigators observed several familial cases of CPA related meningiomas which suggest a strong genetic factor modulating the risk to develop meningiomas in patients who exposed to CPA. The aim of this study is to generate a biobank permitting, in future studies, to identify the genetic locus/loci associated with an increased risk to develop meningiomas after CPA (Androcur®) treatment, using a GWAS approach.

Enrollment of patients will occur at hospitals where the patients will be treated and also via social networking sites such as Facebook. There will be 4 groups of subjects. Five hundred patients will be enrolled in each group targeting 2000 patients in total, among which 1000 patients (Groupe 1 and Groupe 2) will participate in the biobank.

Six centers in 5 university hospitals of APHP (Pitié-Salpêtrière, Ambroise Paré, Cochin, Lariboisière, Saint-Antoine) will be involved in the study.

La duration of enrollment will be 24 months. The participation duration for each subject will be 1 hour. Statistics analysis method: SAS 9.1.3.

ELIGIBILITY:
Inclusion Criteria:

* Age ⩾18 years;
* Non-opposition opinion obtained during the first phone call at the beginning of the study;
* Covered by the french social security scheme.

For the group 1:

* Meningioma diagnosed by medical imaging and confirmed histologically if surgery occurred;
* Cyproterone acetate taken for at least 6 months, 25 mg par day and 20 day by month (cumulated dose ⩾ 3 000mg).

For the group 2:

* Cyproterone acetate taken for at least 5 years with dose of 50 mg per day and 20 day by month, or a cumulated dose corresponding to a longer period (⩾ 30 000mg);
* Normal result of RMI examination performed after at least 5 years treatment by cyproterone acetate.

For the group 3 :

* Subject who has never taken cyproterone acetate;
* Meningioma diagnosed by medical imaging examination and confirmed histologically if surgery occured.

For the group 4 :

* Subject who has never taken cyproterone acetate;
* Subject never diagnosed with meningioma.

Exclusion Criteria:

* Subject under tutoraship;
* Subject refusal;
* Communication difficulties such as: language barriers, serious problems of hearing without a hearing instrument, cognitive troubles... ;
* Foreign subject under AME scheme (a french social system).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Adult women with or without meningioma either exposed or not to cyproterone acetate.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2025-04-19 (Estimated); Study Completion 2025-04-19 (Estimated)

PRIMARY OUTCOMES:
Number of enrolled patients for smear samples | at the end of study, an average of 2 years
  Number of enrolled patients in the study with good quality of smear samples.

SECONDARY OUTCOMES:
Number of family cases of meningioma | at the end of study, an average of 2 years
  Number of family cases of meningioma occurrence will be noted in each group.
Occurrence of meningioma in first-degree relatives | at the end of study, an average of 2 years
  Number of occurrence of meningioma will be collected for:
  * in first-degree relatives of index case in each group.
  * in first-degree relatives exposed to cyproterone acetate in each group.
Occurrence of hormonodependant cancer | at the end of study, an average of 2 years
  Number of hormonodependant cancer occurrence the index case and in first-degree relatives in each group.
Characteristic of the meningioma : Size, Localization, treatment, evolution of meningioma | at baseline
  In goups 1 and 3.
  Size and Localization of meningioma will be determined by RMI examination.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure RAFFIN-SANSON, MD, PhD, Principal Investigator — Service Endocrinologie Nutrition, Hôpital Ambroise Paré, APHP & EA4340, UFR Santé Simone Veil, Université Paris Saclay; Marc SANSON, MD, PhD, Study Chair — Equipe Génétique et Développement des Tumeurs Cérébrales, Service Neuro Oncologie, Hôpital Pitié Salpetrière, APHP
Locations (1):
- Endocrinology Nutrition Department, Ambroise Paré Hospital, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No